CLINICAL TRIAL: NCT04161300
Title: Comparison Between Foam Rolling and Orthopaedic Manual Physical Therapy on Functional Variables in Athletes: A Randomized Controlled Trial
Brief Title: Foam Rolling and Orthopaedic Manual Physical Therapy in Athletes
Acronym: FRvsMTAth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID0027
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Athletic Injuries
MeSH Terms: conditions — Athletic Injuries | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Foam Rolling Group (FR) (Active Comparator)
  Interventions: Other: Foam Rolling (FR)
- Orthopaedic Manual Physical Therapy Group (OMPT) (Active Comparator)
  Interventions: Other: Orthopaedic Manual Physical Therapy Group (OMPT)
- Control Group (CG) (Other)
  Interventions: Other: Control Group (CG)

INTERVENTIONS:
Other: Foam Rolling (FR) — FR auto-massage will place the foam roller between their ischial tuberosity and a hard surface (i.e., the floor) with their legs held in an extended position, keeping their ankles relaxed and oriented upward. For FR in the lumbar region, participants use their weight to slide the FR through the erector of the lumbar and thoracic spine. The total approximate duration will be about 10-15 minutes.
  Arms: Foam Rolling Group (FR)
Other: Control Group (CG) — The CG did not receive any intervention.
  Arms: Control Group (CG)
Other: Orthopaedic Manual Physical Therapy Group (OMPT) — Based on the protocol used by Espí-López et al.: a) Unspecific and bilateral lumbar thrust (L5-S1), one of each side were performed; b) Hip joint decompression, performing 25 repetitions c) Hip rotator stretch with hip and knee flexion, 15 repetitions; d) Femorotibial decompression, 25 reps. e) Quadriceps femoral muscle compression and traction, 25 repetitions; f) Opening of the internal and external femorotibial interline, 15 repetition; g) Ankle decompression, 3 repetitions; h) Posteroanterior and anteroposterior mobilization of head and base of fibula, 25 repetitions. The total duration will be approximately 10-15 minutes.
  Arms: Orthopaedic Manual Physical Therapy Group (OMPT)

SUMMARY:
The main objective of the present study was to evaluate whether FR massage is effective in improving dynamic balance, flexibility and dynamic strength after intense exercise recovery compared to OMPT protocol or a control group. The present study was a randomized controlled trial. Amateur athletes will be recruited from two athletic clubs. Participants will be randomizing and allocating into three non-balanced groups through a computer software by an external assistant who will be blinding to the study objectives: FR group (n = 18), OMPT group (n = 15) and control group (CG) (n = 14). The intervention period will be lasting one day (1 session). Participant assessment will be perform twice: prior to the study (pre-intervention) and immediately after finishing the intervention (post-intervention).

Interventions: FR group. FR auto-massage will place the foam roller between their ischial tuberosity and a hard surface (i.e., the floor) with their legs held in an extended position, keeping their ankles relaxed and oriented upward. For FR in the lumbar region, participants use their weight to slide the FR through the erector of the lumbar and thoracic spine. The total approximate duration will be about 10-15 minutes; OMPT group. Based on the protocol used by Espí-López et al.: a) Unspecific and bilateral lumbar thrust (L5-S1), one of each side were performed; The total duration will be approximately 10-15 minutes.; CG. The CG did not receive any intervention.

Outcomes will be Lumbar flexibility, Hip flexion, Dynamic balance, Standing Jump and Impression of Change.

DETAILED DESCRIPTION:
Introduction Foam rolling (FR) is a form of self-massage in which the targeted musculature is rolled and compressed using a FR. In the field of physical therapy that has been shown to produce a reduced feeling of fatigue in healthy athletes12 as well as hypoalgesic effects in subjects with delayed-onset muscle soreness.

Currently, self-massage through FR is commonly used in the sports field. The reason for this is that it has been suggested that it could have the positive effects traditionally associated with orthopedic manual physical therapy (OMPT), That is why despite the widespread use of FR massage in the field of muscle recovery in athletes, there is a lack of scientific literature about its effectiveness compared to OMPT that can justify its use. Therefore, the main objective of the present study was to evaluate whether FR massage is effective in improving dynamic balance, flexibility and dynamic strength after intense exercise recovery compared to OMPT protocol or a control group.

Methods The present study was a randomized controlled trial. Participants Amateur athletes will be recruited from two athletic clubs. The inclusion criteria will be as follows: (a) male and female amateur athletes aged 18 to 30 years. The exclusion criteria: (a) previous surgery of the locomotor system in lower limbs; (b) musculoskeletal injuries in any part of the body that prevent practicing sports; (c) understanding or communication difficulties; and (d) insufficient fluency in the Spanish language to follow measurement instructions.

Informed written consent will be obtaining from all the participants prior to inclusion. All the participants will be explaining the study procedures, which will be design according to the ethical standards of the Helsinki Declaration.

Procedure Participants will be randomizing and allocating into three non-balanced groups through a computer software by an external assistant who will be blinding to the study objectives: FR group (n = 18), OMPT group (n = 15) and control group (CG) (n = 14). The intervention period will be lasting one day (1 session).

Participant assessment will be perform twice: prior to the study (pre-intervention) and immediately after finishing the intervention (post-intervention).

Interventions FR group. FR auto-massage will place the foam roller between their ischial tuberosity and a hard surface (i.e., the floor) with their legs held in an extended position, keeping their ankles relaxed and oriented upward. For FR in the lumbar region, participants use their weight to slide the FR through the erector of the lumbar and thoracic spine. The total approximate duration will be about 10-15 minutes.

OMPT group. Based on the protocol used by Espí-López et al.: a) Unspecific and bilateral lumbar thrust (L5-S1), one of each side were performed; b) Hip joint decompression, performing 25 repetitions c) Hip rotator stretch with hip and knee flexion, 15 repetitions; d) Femorotibial decompression, 25 reps. e) Quadriceps femoral muscle compression and traction, 25 repetitions; f) Opening of the internal and external femorotibial interline, 15 repetition; g) Ankle decompression, 3 repetitions; h) Posteroanterior and anteroposterior mobilization of head and base of fibula, 25 repetitions. The total duration will be approximately 10-15 minutes.

CG. The CG did not receive any intervention.

Primary outcomes: Physical functional variables Lumbar flexibility. Modified Schober test (MMST). The MMST was designed to assess the mobility of the entire lower back, so the MMST was used to measure lumbar flexion before and after FR and TM interventions. The examiner will place his thumbs on the lower margin of the posterior-upper iliac spine (lower reference point) and a pen mark was made. While the examiner held the tape against the subject's skin, another signal was marked 15 cm above the first (upper reference point). Each subject was then asked to perform an active flexion of the entire trunk and the distance between the two points will be measuring and then the subject return to his initial position. The difference between the initial distance and the new bending measurements will be take.

Hip flexion. by the passive straight leg raise (SLR). Passive SLR will be conducting using a procedure previously described by Hopper et al. A Richards splint and an ankle foot orthosis were applied to the left leg to maintain the knee in full extension and the ankle at a neutral plantar angle. An inclinometer will be attaching to a belt, which will place around the pelvis at the level of the anterior superior iliac spine (Baseline Bubble Inclinometer. Fabrication Enterprises, PO Box, 1500 White Plains, NY 10602, USA). A second inclinometer will be then attaching to the Richards splint at the level of the knee joint line. The mean of 3 measures will be using for analysis. During the test, the participants are positioned with their hands on the abdomen, cervical spine in a neutral position and eyes closed.

Dynamic balance using the Star Excursion Balance Test (SEBT). The SEBT is a dynamic test that requires strength, flexibility, and proprioception. The goal of the SEBT is to maintain single-leg stance while reaching as far as possible with the contralateral leg. Subjects are instructed to stand with both feet positioned inside the boundaries of the starting box. The test initiates when the subject begins to reach in one of the four diagonal directions.

Standing Jump. Subjects are placed their feet shoulder-width apart and toes placed in a line on the floor. The subjects then made a horizontal leap forward, where they were allowed the arms to swing, and it will be done along the length of a tape measure that was fixed to the ground. The subjects had to stick to the ground in the landing phase, preventing any additional movement of the feet when landing.

The jumped distance will be calculating as the distance from the jump initiation line to the heel of the back foot. The best of three attempts was recorded, with a recovery of 60 seconds between attempts. All distances will be measuring with an accuracy of 0.01 meters.

Secondary outcome:

Impression of Change (CGI). Patient Global Impression of Change Scale (PGIOCS) that evaluates the change perceived by the subject after a treatment. This scale has 7 affirmations to choose from (I have improved a lot, quite, a little, I am the same, I have worsened a little, a lot or a lot) and a pain analogue scale of 10 cm.

ELIGIBILITY:
Inclusion Criteria:

* male and female amateur athletes

Exclusion Criteria:

* previous surgery of the locomotor system in lower limbs
* musculoskeletal injuries in any part of the body that prevent practicing sports understanding or communication difficulties
* insufficient fluency in the Spanish language to follow measurement instructions.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Dynamic balance | 1 day
  Dynamic balance using the Star Excursion Balance Test (SEBT). The SEBT is a dynamic test that requires strength, flexibility, and proprioception. The goal of the SEBT is to maintain single-leg stance while reaching as far as possible with the contralateral leg. Subjects are instructed to stand with both feet positioned inside the boundaries of the starting box. The test initiates when the subject begins to reach in one of the four diagonal directions.

SECONDARY OUTCOMES:
Perception of Change | 1 day
  Patient Global Impression of Change Scale (PGIOCS) that evaluates the change perceived by the subject after a treatment. This scale has 7 levels which represent improvement from 1 to 3, 4 indicates no change and 5 to 7 indicates worsening. In addition, it includes a visual analog scale which scores range from 0 to 10 where 0 is much better and 10 much worse.
Lumbar flexibility | 1 day
  Modified Schober test (MMST). The MMST was designed to assess the mobility of the entire lower back, so the MMST was used to measure lumbar flexion before and after FR and TM interventions. The examiner will place his thumbs on the lower margin of the posterior-upper iliac spine (lower reference point) and a pen mark was made. While the examiner held the tape against the subject's skin, another signal was marked 15 cm above the first (upper reference point). Each subject was then asked to perform an active flexion of the entire trunk and the distance between the two points will be measuring and then the subject return to his initial position. The difference between the initial distance and the new bending measurements will be take.
Hip flexion | 1 day
  Hip flexion by the passive straight leg raise (SLR). Passive SLR will be conducting using a procedure previously described by Hopper et al. A Richards splint and an ankle foot orthosis were applied to the left leg to maintain the knee in full extension and the ankle at a neutral plantar angle. An inclinometer will be attaching to a belt, which will place around the pelvis at the level of the anterior superior iliac spine (Baseline Bubble Inclinometer. Fabrication Enterprises, PO Box, 1500 White Plains, NY 10602, USA). A second inclinometer will be then attaching to the Richards splint at the level of the knee joint line. The mean of 3 measures will be using for analysis. During the test, the participants are positioned with their hands on the abdomen, cervical spine in a neutral position and eyes closed.
Standing Jump | 1 day
  Subjects are placed their feet shoulder-width apart and toes placed in a line on the floor. The subjects then made a horizontal leap forward, where they were allowed the arms to swing, and it will be done along the length of a tape measure that was fixed to the ground. The subjects had to stick to the ground in the landing phase, preventing any additional movement of the feet when landing.
  The jumped distance will be calculating as the distance from the jump initiation line to the heel of the back foot. The best of three attempts was recorded, with a recovery of 60 seconds between attempts. All distances will be measuring with an accuracy of 0.01 meters.

CONTACTS AND LOCATIONS:
Overall Officials: Gemma V Espí-López, Dr, Principal Investigator — Faculty of Physiotherapy. University of Valencia
Locations (1):
- Gemma v. Espí López, Valencia, Spain

REFERENCES:
- [Derived] Espi-Lopez GV, Ruescas-Nicolau MA, Castellet-Garcia M, Suso-Marti L, Cuenca-Martinez F, Marques-Sule E. Effectiveness of Foam Rolling vs. Manual Therapy in Postexercise Recovery Interventions for Athletes: A Randomized Controlled Trial. J Strength Cond Res. 2023 Jun 1;37(6):e361-e368. doi: 10.1519/JSC.0000000000004383. Epub 2022 Dec 19. PMID 36534492